CLINICAL TRIAL: NCT04437654
Title: The Efficacy and Safety of Non-vItamiN K antaGonist oraL Anticoagulants for intermEdiate Stroke Risk in Patients With Atrial Fibrillation (SINGLE-AF)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0438
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation Patients With Intermediate Stroke Risk
Keywords: Atrial fibrillation; anticoagulation; intermediate stroke risk; efficacy; safety
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anticoagulation group(Apixaban group) (Experimental): Apixaban 5mg twice daily (2.5mg twice daily if meets dose-reduction criteria) for 2 years
  Interventions: Drug: Anticoagulation group(Apixaban group)
- Nonanticoagulation group (No Intervention): Standard treatment except anticoagulant for 2 years

INTERVENTIONS:
Drug: Anticoagulation group(Apixaban group) — Apixaban 5mg twice daily (2.5mg twice daily if meets dose-reduction criteria) for 2 years
  Arms: Anticoagulation group(Apixaban group)

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of non-vitamin K antagonist oral anticoagulants (NOAC) in atrial fibrillation patients with intermediate stroke risk (CHA2DS2-VASc score 1 for male, 2 for female).

A. Major safety results include major bleeding and clinically relevant non-major bleeding.

B. Major efficacy results include strokes, systemic embolism and cardiovascular mortality.

C. Other results include myocardial infarction, pulmonary embolism, transient ischemic attack, hospitalization, drug compliance, quality of life questionnaire (AFEQT), cognitive function (KDSQ), aging questionnaire(K-Frail) and hand grip strength.

ELIGIBILITY:
Inclusion Criteria:

* Age: 19~80 years old
* CHA2DS2-VASc score 1 for male or 2 for female among nonvalvular atrial fibrillation patients
* Patients who agree to register for this study
* Patients who can be observed for the progress after treatment

Exclusion Criteria:

* Severe liver or kidney dysfunction
* Thyroid dysfunction
* Pregnant or breastfeeding women
* Malignant tumors that have not been completely cured
* Severe structural heart disease
* Predicted survival is less than 12 months
* Patients who do not understand the content of the study or disagree with it

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — CHA2DS2-VASc score 1 for male, 2 for female.
Enrollment: 1800 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | Baseline
  Composite outcome including stroke/systemic embolism, major bleeding, and cardiovascular death
Composite outcome | 1 month
  Composite outcome including stroke/systemic embolism, major bleeding, and cardiovascular death
Composite outcome | 6 months
  Composite outcome including stroke/systemic embolism, major bleeding, and cardiovascular death
Composite outcome | 12 months
  Composite outcome including stroke/systemic embolism, major bleeding, and cardiovascular death
Composite outcome | 18 months
  Composite outcome including stroke/systemic embolism, major bleeding, and cardiovascular death
Composite outcome | 24 months
  Composite outcome including stroke/systemic embolism, major bleeding, and cardiovascular death

SECONDARY OUTCOMES:
Stroke | Baseline
  )Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Stroke | 1 month
  )Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Stroke | 6 months
  )Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Stroke | 12 months
  )Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Stroke | 18 months
  )Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Stroke | 24 months
  )Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Systemic embolism | Baseline
  Systemic embolism refers to emboli in the arterial circulation, and defined by both clinical and objective evidence of sudden loss of end-organ perfusion.
Systemic embolism | 1 month
  Systemic embolism refers to emboli in the arterial circulation, and defined by both clinical and objective evidence of sudden loss of end-organ perfusion.
Systemic embolism | 6 months
  Systemic embolism refers to emboli in the arterial circulation, and defined by both clinical and objective evidence of sudden loss of end-organ perfusion.
Systemic embolism | 12 months
  Systemic embolism refers to emboli in the arterial circulation, and defined by both clinical and objective evidence of sudden loss of end-organ perfusion.
Systemic embolism | 18 months
  Systemic embolism refers to emboli in the arterial circulation, and defined by both clinical and objective evidence of sudden loss of end-organ perfusion.
Systemic embolism | 24 months
  Systemic embolism refers to emboli in the arterial circulation, and defined by both clinical and objective evidence of sudden loss of end-organ perfusion.
Major bleeding | Baseline
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Major bleeding | 1 month
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Major bleeding | 6 months
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Major bleeding | 12 months
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Major bleeding | 18 months
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Major bleeding | 24 months
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Clinically Relivant Non-Major Bleeding (CRNMB) | Baseline, 1month, 6 month, 12 month, 18 month, 24 month
  1. Any sign or symptom of hemorrhage (e.g., more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria: i. requiring medical intervention by a healthcare professional ii. leading to hospitalization or increased level of care iii. prompting a face to face (i.e., not just a telephone or electronic communication) evaluation 2. ISTH major bleeding in non-surgical patients is defined as having a symptomatic presentation and 1: i. Fatal bleeding, and/or ii. Bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or iii. Bleeding causing a fall in hemoglobin level of 20 g L-1 (1.24 mmol L-1) or more, or leading to transfusion of two or more units of whole blood or red cells.
Death | Baseline, 1month, 6 month, 12 month, 18 month, 24 month
  the permanent stopping of all the vital bodily activities
Transient ischemic attack (TIA) | Baseline, 1month, 6 month, 12 month, 18 month, 24 month
  TIA is brief episodes of neurological dysfunction resulting from focal cerebral ischemia not associated with permanent cerebral infarction.
Hospital admission | Baseline, 1month, 6 month, 12 month, 18 month, 24 month
  Hospital admission means admission of a covered person to a hospital as an inpatient for medically necessary and appropriate care and treatment of an Illness or Injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No